CLINICAL TRIAL: NCT02240173
Title: Phase 2 Study of the Antipsychotic Effects of Sorghum Bicolor (JOBELYN) in the Treatment of Schizophrenia.
Brief Title: Antipsychotic Effects of Sorghum Bicolor (JOBELYN) in the Treatment of Schizophrenia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal Neuro-Psychiatric Hospital, Yaba (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MOjo
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Schizophrenia and Disorders With Psychotic Features
Keywords: antipsychotic Jobelyn schizophrenia sorghum bicolor
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Haloperidol; haloperidol decanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jobelyn + Haloperidol (Experimental): Combination of the conventional drugs and Jobelyn
  Interventions: Dietary Supplement: Jobelyn
- Haloperidol + Placebo (Active Comparator): Combination of the conventional drug + Placebo
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Dietary Supplement: Jobelyn — Jobelyn is a dietary supplement made from Sorghum bicolor
  Other Names: Sorghum bicolor
  Arms: Jobelyn + Haloperidol
Drug: Haloperidol — Conventional drug normally used for psychotic problems
  Other Names: Haloperidol decanoate
  Arms: Haloperidol + Placebo

SUMMARY:
Sorghum bicolor is a naturally growing plant which has been of health benefit to the people of West Africa who traditionally prepare its leaf for various nutritional and health reasons.The food and nutritional fact analysis showed that Jobelyn is rich in Carbohydrates, Protein, Dietary Fiber, Iron, Natural Vitamins like B12 and Vitamin C. It also contains Selenium, Omega 3,6 and 9 and other essential elements and fatty acids. Although the determinants of mental health are complex, the emerging and compelling evidence for nutrition as a crucial factor in the high prevalence and incidence of mental disorders suggests that diet is as important to psychiatry as it is to cardiology, endocrinology, and gastroenterology. Evidence is steadily growing for the relation between dietary quality (and potential nutritional deficiencies) and mental health, and for the select use of nutrient-based supplements to address deficiencies, or as monotherapies or augmentation therapies. There is currently strong advocacy for the recognition of diet and nutrition as central determinants of both physical and mental health.Its anti-inflammatory and haematocrit boosting properties have been well documented though the precise mechanism of action is still largely unknown. Its use has recently been extended to the field of mental health where findings in animal study suggest it could be of help in relieve of psychosis. The need for this study is therefore aimed at investigating the effect of this drug in patients with schizophrenia which is the prototypical psychotic disorder.

DETAILED DESCRIPTION:
Schizophrenia is a major psychiatric disorder with a chronic and debilitating course. It is the archetypal psychotic disorder with a prevalence of about 1% worldwide. The treatment of this psychotic disorder has evolved over the years after the discovery of Chlorpromazine. Despite the availability of several treatment options in practice, research into the possibility of creating a drug breakthrough continues.

Sorghum bicolor, a naturally growing plant rich in several phytochemical including proanthocyanidins, anthocyanidins, apigenin, proapigeninidin, apigeninidin, luteolin, naringenins, flavonoids, and polyphenols (Omogbiya et al 2012) and prepared as a capsule called Jobelyn. This plant has been found to be of health benefit to the people of West Africa who traditionally prepare its leaf for various nutritional and health reasons. The anti-inflammatory and haematocrit boosting properties have been well documented and utilized though the precise mechanism of action is still not entirely known (Benson et al. 2013). Its usefulness in neuropsychiatric conditions has recently been explored albeit through animal studies.

In animals, Jobelyn has been suggested to have anti-amnestic property which has been suggested to be related to its antioxidant activity (Umukoro et al. 2013a). Other studies also suggested that Jobelyn has an anti-aggressive effect (Umukoro et al. 2012) and antidepressant like property probably related to its stimulation of serotonergic pathways (Umukoro et al. 2013b). Jobelyn has also been suggested to exhibit anti-psychotic-like activity with the benefit of lacking extra-pyramidal side effect risks and therefore being postulated to be of possible benefit in the symptomatic relief of psychosis (Omogbiya et al. 2012).

There is however limited information in terms of the suggested neuropsychiatric conditions especially in humans despite the recognized safety profile consequent upon its use as haematocrit boosting agent. This study therefore aims at exploring the usefulness of Jobelyn in the treatment of patients with Schizophrenia as an adjunct to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants will be adults with current diagnosis of schizophrenia (meeting the ICD-10 criteria).

* Adults who are above 18 years of age and gave informed consent
* Currently meet the ICD-10 diagnosis of Schizophrenia and confirmed with MINI- PLUS
* Antipsychotic naive before recruitment into study or defaulted from treatment for at least 6 months 'prior to contact with study
* Not on Jobelyn or Megafit currently or in the past 6months prior to contact with study

Exclusion Criteria:

* Having another current ICD-l0 diagnosis or a seizure disorder
* Serious or chronic physical illness
* Known severe drug allergies or hypersensitivity to Jobelyn, Megafit or Haloperidol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the changes in psychotic symptoms | 8 Weeks
  This will be rated using the Brief Psychiatric Rating Scale (BPRS).

SECONDARY OUTCOMES:
Patient's general health and social functioning | 8 Weeks
  To be assessed using the Clinical Global Impression Scale.

OTHER OUTCOMES:
Side effects | 8 Weeks
  This will be measured using a side-effect scale designed for the study

CONTACTS AND LOCATIONS:
Overall Officials: Moses Ojo, M.D., Principal Investigator — NPHY
Locations (1):
- Federal Neuro-Psychiatric Hospital Yaba - Lagos, Lagos, Lagos, Nigeria

REFERENCES:
- [Background] Ayuba GI, Jensen GS, Benson KF, Okubena AM, Okubena O. Clinical efficacy of a West African sorghum bicolor-based traditional herbal preparation Jobelyn shows increased hemoglobin and CD4+ T-lymphocyte counts in HIV-positive patients. J Altern Complement Med. 2014 Jan;20(1):53-6. doi: 10.1089/acm.2013.0125. Epub 2013 Nov 27. PMID 24283768
- [Background] Geera B, Ojwang LO, Awika JM. New highly stable dimeric 3-deoxyanthocyanidin pigments from sorghum bicolor leaf sheath. J Food Sci. 2012 May;77(5):C566-72. doi: 10.1111/j.1750-3841.2012.02668.x. Epub 2012 Apr 10. PMID 22489620
- [Background] Benson KF, Beaman JL, Ou B, Okubena A, Okubena O, Jensen GS. West African Sorghum bicolor leaf sheaths have anti-inflammatory and immune-modulating properties in vitro. J Med Food. 2013 Mar;16(3):230-8. doi: 10.1089/jmf.2012.0214. Epub 2013 Jan 5. PMID 23289787
- [Background] Umukoro S, Omogbiya IA, Eduviere AT. Evaluation of the effect of jobelyn((R)) on chemoconvulsants-induced seizure in mice. Basic Clin Neurosci. 2013 Spring;4(2):125-9. PMID 25337338
- [Background] Umukoro S, Ugbomah A, Aderibigbe A, Omogbiya A. Antioxidant Property of Jobelyn as the Possible Mechanism Underlying its Anti-amnesic Activity in Rodents. Basic Clin Neurosci. 2013 Winter;4(1):42-9. PMID 25337327
- [Background] Omogbiya IA, Umukoro S, Aderibigbe AO, Bakre AG. Jobelyn(R) pretreatment ameliorates symptoms of psychosis in experimental models. J Basic Clin Physiol Pharmacol. 2013;24(4):331-6. doi: 10.1515/jbcpp-2012-0073. PMID 23412872
- [Background] Umukoro S, Omogbiya IA, Eduviere TA. Effect of Jobelyn(R) on intruder- and isolation-induced aggressive behavior in mice. J Basic Clin Physiol Pharmacol. 2013;24(4):263-9. doi: 10.1515/jbcpp-2012-0069. PMID 23729562
- [Background] Toxicological Profiles of Commercial Herbal Preparation, Jobelyn® nternational Journal of Health Research, December 2009; 2(4): 369-374 © Poracom Academic Publishers. All rights reserved. Available at http://www.ijhr.org
- [Background] The influence of African Herbal Formula on the haematological parameters of trypanosome infected rats VI Okochi, J Okpuzor, MO Okubena, AK Awoyemi African Journal of Biotechnology Vol.2(9) 2003: 312-316
- [Background] Response of Trypanosoma brucei brucei-induced anaemia to a commercial herbal preparation ........... 4 African Journal of Biotechnology Vol. 2 (9), pp. 307-311, September 2003
- [Background] Yang L, Dykes L, Awika JM. Thermal stability of 3-deoxyanthocyanidin pigments. Food Chem. 2014 Oct 1;160:246-54. doi: 10.1016/j.foodchem.2014.03.105. Epub 2014 Apr 1. PMID 24799235